CLINICAL TRIAL: NCT01344798
Title: Phase I Clinical Study of AAV1-gamma-sarcoglycan Gene Therapy for Limb Girdle Muscular Dystrophy Type 2C
Brief Title: Clinical Study of AAV1-gamma-sarcoglycan Gene Therapy for Limb Girdle Muscular Dystrophy Type 2C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genethon (Other)
Responsible Party: Frederic Revah, CEO, Genethon
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTG001.06
Record Dates: First submitted 2011-03-17; First posted 2011-04-29 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Limb Girdle Muscular Dystrophy Type 2C; Gamma-sarcoglycanopathy
Keywords: limb girdle muscular dystrophy type 2C; gamma-sarcoglycanopathy; gene therapy; AAV vector; neuromuscular disease; orphan disease
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 2C; Neuromuscular Diseases; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose level 1 (Experimental): AAV1-gamma-sarcoglycan vector dose level: 3x10e9 vg/100µl
  Interventions: Biological: AAV1-gamma-sarcoglycan vector injection
- Dose level 2 (Experimental): AAV1-gamma-sarcoglycan vector dose level: 1.5x10e10 vg/100µl
  Interventions: Biological: AAV1-gamma-sarcoglycan vector injection
- Dose level 3 (Experimental): AAV1-gamma-sarcoglycan vector dose level: 4.5x10e10 vg/300µl
  Interventions: Biological: AAV1-gamma-sarcoglycan vector injection

INTERVENTIONS:
Biological: AAV1-gamma-sarcoglycan vector injection — single intramuscular injection into carpi radialis muscle under open procedure
  Other Names: in vivo gene therapy - Intramuscular route

SUMMARY:
The purpose of this trial is to study the evaluation of clinical safety and feasibility of gene therapy in patients with limb girdle muscular dystrophy type 2C (gamma-sarcoglycanopathy).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of LGMD 2C including:

   * Molecular analysis proving del525T mutation on γ-sarcoglycan gene (chromosome 13) at homozygous state
   * Muscle biopsy with immunohistochemical and/or Western blot analyses showing marked decrease or absence of γ-sarcoglycan staining in muscle, as well as a fibrosis assessment should be available. If not, an initial muscular biopsy may be performed during the pre-enrollment period
2. Lower age limit of 15 years
3. Males and females may be equally enrolled
4. Adequate carpi radialis muscle bulk for muscle biopsy as assessed by examination. Subjects should be able to communicate with the investigation staff. They should be able to understand, to comply with and to perform all needed evaluations during the trial period, including muscle strength tests. Forearm muscle strength should be of at least 3+ as assessed through the British Medical Research Council (MRC) Manual Muscle Testing (MMT) scale.

   Subjects should also have already lost ambulation
5. Subjects should be able and willing to return for follow up
6. Subjects should be able and willing to give signed informed consent. For minor subjects, a signed informed consent will be given by legally authorized representative
7. Eligible subjects belonging to a multiplex family should not be enrolled in the same cohort.

Exclusion Criteria:

1. Severity of disease and presence of ill-prognosis complications:

   * Severe respiratory dysfunction such as subjects with tracheostomy or forced vital capacity (FVC) < 1000 ml and/or < 30%;
   * Uncompensated heart failure;
   * An ejection fraction (EF) < 30% as measured on either echocardiography or scintigraphy;
   * Severe rhythm disturbances and/or high degree conduction defect in the absence of a pacemaker insertion.
2. Underlying conditions, diseases or active viral infections likely to increase risk of complications or to interfere with the investigational treatment:

   * contraindications for injections and muscle biopsies
   * Platelet count < 100,000 / mm3
   * Total bilirubin > 10 mg/l (> 17 µmol/l)
   * Serum creatinin > 110 µmol/l
   * Lymphocytes CD4+ < 250/mm3 (< 15%)
   * History of diabetes mellitus
   * Current infectious diseases, including known positive HIV serology, hepatitis B and C
   * Abnormal profile on protein immunoelectrophoresis
   * Immunizations of any kind within the past month
   * receipt of another investigational agent within 4 weeks of study enrollment
   * History of or current steroid medication for indications other than muscular dystrophy, chemotherapy, radiotherapy or other immunosuppressive therapy. Steroid medication, if any, should be discontinued at least 3 months before entering the protocol and not received during the study
   * Pregnant or lactating women. Females or males of childbearing age must be willing to employ adequate contraception, that is to use condoms during the 3 months following the administration of the product
   * Pre-injection neutralizing anti-AAV1 antibodies titer (on pre-enrollment / D-30 visit) superior or equal to 1/800.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events or general or local signs as a measure of clinical safety | 6 months
  Standard general and local clinical examination as well as vital signs assessement, including pain, local inflammation, stiffness and fatigability.

SECONDARY OUTCOMES:
Number of patients with modified biological values (blood count, standard biochemistry, viral serology) | 6 months
  Assessment of biological tolerance:
  * blood count
  * standard biochemistry
  * CPK viral serology (hepatitis B & C)
number of patients with changed or increased humoral immunity to AAV | 6 months
  assessment of anti-AAV antibodies titers
Number of patients with changed/increased humoral immunity to transgene | 6 months
  assessment of anti-gamma-sarcoglycan antibodies titers
Number of patients with changed/increased cellular immunity to AAV | 6 months
  assessment cellular immunity against AAV (ELispot assay)
Number of patients with changed/increased cellular immunity to transgene | 6 months
  assessment cellular immunity against gamma-sarcoglycan (ELispot assay)
number of patients with positively stained muscular fibers to gamma-sarcoglycan protein | 30 days
  Muscular biopsy immunohistaining for the detection of gamma-sarcoglycan
Number of patients with modified/decreased muscular force | 6 months
  functional testing of treated muscle through a specially designed ergometer

CONTACTS AND LOCATIONS:
Overall Officials: Serge Herson, Prof, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France